CLINICAL TRIAL: NCT03744364
Title: Low-dose Vaginal Misoprostol Versus Vaginal Dinoprostone Insert for Induction of Labor Beyond 41st Week: a Randomized Trial
Brief Title: Low-dose Vaginal Misoprostol Versus Vaginal Dinoprostone Insert for Induction of Labor
Acronym: MADUTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Jose Manuel Campillos Maza, Head of Unit of Maternal-Fetal Medicine, Hospital Miguel Servet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JMC-PGE-2014-01
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Induced Labor; Cervical Ripening; Obstetric Labor; Pregnancy
Keywords: Dinoprostone; Misoprostol
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol (Active Comparator): Group of women allocated to misoprostol induction.
  Interventions: Drug: Misoprostol 25 mcg
- Dinoprostone (Active Comparator): Group of women allocated to dinoprostone induction.
  Interventions: Drug: Dinoprostone 10mg

INTERVENTIONS:
Drug: Misoprostol 25 mcg — To determine efficacy and safety of vaginal 'Misoprostol 25 mcg' every 4 hours with a maximum of 6 doses for induction of labor.
  Other Names: Misoprostol induction
  Arms: Misoprostol
Drug: Dinoprostone 10mg — To determine efficacy and safety of 'Dinoprostone 10mg' vaginal insert for induction of labor.
  Other Names: Dinoprostone induction
  Arms: Dinoprostone

SUMMARY:
Purpose:

To compare the efficacy and safety of low-dose protocol of vaginal misoprostol and vaginal dinoprostone insert for induction of labor in women with post-term pregnancies.

Methods:

The investigators designed a prospective, randomized, open-labeled, blinded for the end-point evaluators trial including women of at least 41 weeks of gestational age with uncomplicated singleton pregnancies and Bishop score lower than 6. Participants were randomized into dinoprostone or misoprostol groups in a 1:1 ratio. Baseline maternal data and perinatal outcomes were recorded for statistical analysis. Successful vaginal delivery within 24 hours was the primary outcome variable.

ELIGIBILITY:
Inclusion Criteria:

* Singleton uncomplicated pregnancy
* Nulliparity
* Live fetus
* 286 days of gestational age or above
* Abscence of contraindication for vaginal delivery
* Bishop score lower than 6

Exclusion Criteria:

* Multiple pregnancy
* Multiparity
* Stillbirth
* Oligohydramnios
* Suspected fetal distress
* Severe asthma
* Intolerance/allergy to prostaglandins
* Contraindication for vaginal birth

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 198 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Successful vaginal delivery within 24 hours | 24 hours since induction was started
  Percentage of women that achieve a vaginal delivery within 24 hours since induction process started

SECONDARY OUTCOMES:
Successful cervical ripening within 24 hours | 24 hours since induction was started
  Percentage of women that achieve Bishop score > 6 within 24 hours since induction process started
Interval time from induction to delivery | Hours passed between induction of labor until delivery within 72 hours
  Time passed since induction of labor started until delivery
Need for a second induction | Assessed 24 hours since induction of labor was started
  Percentage of women that require to use a second method for induction of labor after 24 hours of having started induction of labor
Vaginal delivery rate | Since labor induction had started until delivery had ocurred within 72 hours
  Percentage of women that achieve vaginal delivery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Bonrostro Torralba C, Tejero Cabrejas EL, Envid Lazaro BM, Franco Royo MJ, Roca Arquillue M, Campillos Maza JM. Low-dose vaginal misoprostol vs vaginal dinoprostone insert for induction of labor beyond 41st week: A randomized trial. Acta Obstet Gynecol Scand. 2019 Jul;98(7):913-919. doi: 10.1111/aogs.13556. Epub 2019 Feb 24. PMID 30723912